CLINICAL TRIAL: NCT06712082
Title: A Phase 1, Randomized, Double-Blind, Third-Party Open, Placebo-Controlled, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, Tolerability, Immunogenicity, and Pharmacodynamics Following Intravenous Dose of PF-07264660 in Chinese Healthy Adult Participants
Brief Title: A Study to Learn More About the Study Medicine PF-07264660 in Healthy Chinese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: C4521003
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PF-07264660 (Experimental): Participants will receive a single dose of PF-07264660 via IV infusion
  Interventions: Drug: PF-07264660
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo via IV infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-07264660 — PF-07264660 solution for injection (single use only)
  Arms: PF-07264660
Other: Placebo — Placebo solution for injection (single use only)
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn if the study medicine (called PF-07264660) is safe and how it is processed in healthy Chinese participants. This study is seeking participants who:

* are between 18 to 65 years of age.
* are Chinese participants who are overtly healthy as determined by medical evaluation.
* have a BMI (body mass index) of 19 to 28 kilogram per meter squared; and a total body weight of more than50 kilograms (110 pounds).

All participants in this study will receive study medicine. Three-fourths will receive PF-07264660 and one-fourth will receive placebo. A placebo does not have any medicine in it but looks just like the medicine being studied. The study medicine will be given as an IV infusion (directly into a vein) at the study clinic only one time.

The study will compare the experiences of people receiving PF-07264660 to those of people who do not. This will help see if PF-07264660 is safe and how it behaves inside the human body.

Participants will take part in this study for up to 181 days. During this time, the participants will stay at the study clinic for 5 days. After the stay, the participants will have 8 study visits at the study clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants aged 18 to 65 years.
2. Body mass index (BMI) of 19-27.9 kilogram per meter squared, inclusive, and a total body weight >50 kilograms (110 pounds).
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
4. Capable of giving signed informed consent.

Key Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
2. History of human immunodeficiency virus (HIV) infection, hepatitis B, hepatitis C, or syphilis; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb), or syphilis.
3. Evidence of active, latent, untreated or inadequately treated infection with Mycobacterium tuberculosis (TB).
4. Participants with any acute or chronic infections or infection history as per protocol required.
5. History of fever within 7 days prior to dosing.
6. Recent exposure to live or attenuated vaccines within 28 days of the screening visit.
7. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Use of prohibited concomitant medication within 7 days or 5 half-lives (whichever is longer) prior to the administration of PF-07264660.
9. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the administration of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
10. A positive urine drug test.
11. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) following at least 5 minutes of supine rest.
12. Standard 12 lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
13. Participants with any protocol defined abnormalities in clinical laboratory tests at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to Day 181
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to Day181
area under the concentration-time curve from time 0 to 336 hours (AUC336) | Up to Day 181
area under the concentration-time curve from time 0 to infinity (AUCinf) | Up to Day 181
area under the concentration-time curve from 0 to time of last measurable concentration (AUClast) | Up to Day 181
Terminal phase half-life (t½) | Up to Day 181
Incidence of treatment-emergent adverse events (TEAEs) | Up to Day 181
Incidence of treatment-emergent serious adverse events (SAEs) | Up to Day 181
Incidence of abnormal and clinically relevant changes in vital signs | Up to Day 181
Incidence of abnormal and clinically relevant changes in electrocardiogram | Up to Day 181
Incidence of abnormal and clinically relevant changes in laboratory assessments | Up to Day 181

SECONDARY OUTCOMES:
Clearance (CL) of PF-07264660 | Up to Day 181
volume of distribution (Vss) | Up to Day 181
mean residence time (MRT) | Up to Day 181
Incidence of the Development of Anti-Drug Antibodies (ADA) against PF-07264660 | Up to Day 181
Incidence of the neutralizing antibodies (NAb) against PF-07264660, if appropriate and feasible | Up to Day 181
Change from baseline in serum levels of chemokine (C-C motif) ligand 17 (CCL17) / thymus and activation regulated chemokine (TARC) | Up to Day 181
Change from baseline in serum levels of total immunoglobulin E (IgE) | Up to Day 181

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Huashan Hospital,Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4521003